CLINICAL TRIAL: NCT05533567
Title: Electroencephalographic Profiles During General Anesthesia: a Comparative Study of Remimazolam and Propofol
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital of Nanchang University (Other)
Responsible Party: Principal Investigator, Fuzhou Hua, Chief Physician, Second Affiliated Hospital of Nanchang University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2022-EEG-1
Record Dates: First submitted 2022-09-02; First posted 2022-09-09 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: General Anesthesia; Electroencephalography; Laparoscopic Cholecystectomy; Remimazolam; Propofol
Keywords: Electroencephalography; General Anesthesia; Remimazolam; Propofol; Laparoscopic Cholecystectomy
MeSH Terms: interventions — remimazolam; Sufentanil; cisatracurium; Propofol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remimazolam group (Experimental): 1. Induction of anesthesia Slowly injects remimazolam 0.4-0.6 mg/kg (about 1 minute) until loss of consciousness (LoC), if the degree of sedation is insufficient, additional remimazolam (0.05 mg/kg each time) is allowed. After the LoC, intravenous sufentanil 0.3 ~0.5ug/kg and cisatracurium besylate 0.1 mg/kg are injected intravenously. After the muscles are sufficiently relaxed and blood circulation is stable, the tracheal tube is inserted under a glide scope.
  2. Maintenance of anesthesia remimazolam 0.4~1.2 mg/kg/h and remifentanil 0.1~0.3 ug/kg/min are injected intravenously to maintain sedation and assistant analgesia, and cisatracurium besylate 0.02 mg/kg is allowed to add as appropriate. During the operation, the dose of anesthetic drugs is adjusted so that the fluctuation of heart rate and blood pressure did not exceed 10 %.
  Interventions: Drug: Remimazolam
- Propofol group (Active Comparator): 1. Induction of anesthesia Slowly injects propofol 2-4 mg/kg (about 1 min) until loss of consciousness (LoC), allowing additional propofol (0.5 mg/kg each time) if sedation is insufficient. after LoC, intravenous sufentanil 0.3 ~0.5ug/kg and cisatracurium besylate 0.1 mg/kg. after sufficient muscle relaxation and blood circulation stabilization, the tracheal tube was inserted under the sliding scope.
  2. Maintenance of anesthesia propofol 4~10mg/kg/h and remifentanil 0.1~0.3 ug/kg/min are injected intravenously to maintain sedation and assistant analgesia, and cisatracurium besylate 0.02 mg/kg is allowed to add as appropriate. During the operation, the dose of anesthetic drugs is adjusted so that the fluctuation of heart rate and blood pressure did not exceed 10 %.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Remimazolam — The experimental group was sedated with remimazolam.
  Other Names: sufentanil; cisatracurium besylate
  Arms: Remimazolam group
Drug: Propofol — The control group was sedated with propofol.
  Other Names: sufentanil; cisatracurium besylate
  Arms: Propofol group

SUMMARY:
How anesthetic drugs induce and maintain the behavioral state of general anesthesia is an important question in medicine and neuroscience. Different anesthetic drugs act on different molecular targets and neural circuit mechanisms, exhibiting drug-specific EEG features. As a novel ultra-short-acting benzodiazepines drugs, remimazolam has been accepted for induction and maintenance of clinical anesthesia. Compared to the traditional benzodiazepines drugs, remimazolam combines the safety of midazolam with the effectiveness of propofol, and also has the advantages of acting quickly, short half-life, no injection pain, slight respiratory depression, independent of liver and kidney metabolism, long-term infusion without accumulation, and has a specific antagonist: flumazenil. This study aimed to investigate the differences in the characteristics of EEG oscillations during general anesthesia by comparing propofol and remimazolam.

ELIGIBILITY:
Inclusion Criteria:

1. Right-handed, age 18-60 years, sex not limited.
2. Patients proposed to undergo elective laparoscopic cholecystectomy under general anesthesia in the morning, with an expected operative duration of approximately 1h to 2h.
3. Body mass index (BMI) <28 kg/m2.
4. Anxiety score >50, both without anxiety and sleep disorders.
5. ASA anesthesia classification grade I with Mallampati class I airway anatomy.
6. Can communicate effectively with the physician.
7. Patients were aware of and voluntarily signed the informed consent form.

Exclusion Criteria:

1. Relative contraindications to general anesthesia: patients with severe cardiac or pulmonary function disease.
2. Patients taking drugs that may confound EEG or behavioral findings or during pregnancy.
3. Patients with a history of psychiatric or neurological disorders, drug abuse, or drug addiction.
4. Any cerebrovascular accident within 3 months, such as stroke, transient ischemic attack (TIA), etc.;
5. Inability to cooperate in completing the test, or refusal of the patient or family members to participate.
6. Those with known allergies, or allergies to the test drug.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
EEG waveforms | Duration from the time the patient enters the operating room to the time they leave the post-anesthesia care unit, average two hours.
  Contrasting differences in electroencephalographic oscillatory characteristics during general anesthesia with propofol and remimazolam.

SECONDARY OUTCOMES:
systolic pressure | Up to 5 hours including preoperative, intraoperative, and postoperative periods
  Indicators related to perioperative hemodynamics
diastolic pressure | Up to 5 hours including preoperative, intraoperative, and postoperative periods
  Indicators related to perioperative hemodynamics
mean pressure | Up to 5 hours including preoperative, intraoperative, and postoperative periods
  Indicators related to perioperative hemodynamics
heart rate | Up to 5 hours including preoperative, intraoperative, and postoperative periods
  Indicators related to perioperative hemodynamics
pulse | Up to 5 hours including preoperative, intraoperative, and postoperative periods
  Indicators related to perioperative hemodynamics
Recovery times | Up to 30 minutes after operation
  The period from discontinuation of anesthetic drugs to the recovery of the patient's self-consciousness and can respond correctly to external stimuli. All the patients can be allowed to leave the post-anesthesia care unit after Aldrete ≥ 9. Delayed awakening is defined as failure to achieve Aldrete ≥ 9 more than 30 minutes after surgery.
Complication | During the perioperative period
  All the perioperative complications are recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- the Second Affiliated Hospital of Nanchang University, Nanchang University, Nanchang, Jiangxi, China